CLINICAL TRIAL: NCT05197634
Title: The Impact of Covid-19 Pandemic, On The Eating Habits, Lifestyle Changes and Traumatic Injuries In The Children With Autism Spectrum Disorder
Brief Title: The Impact of Covid-19 Pandemic On The Children With Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: Istanbul Kent University (Other)
Responsible Party: Principal Investigator, Yelda Kasımoğlu, Principal investigator, Istanbul University
Other Study IDs: 2021/49
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Autism With High Cognitive Abilities; COVID-19 Pandemic
Keywords: ASD (autism spectrum disorder); Covid-19; Dental trauma; Eating habits; Lifestyle changes
MeSH Terms: conditions — COVID-19; Autism Spectrum Disorder; Feeding Behavior | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Autism Spectrum Disorder: The orofacial trauma history, dietary habits and lifestyle changes of children aged 3-14 years diagnosed with autism in Istanbul University Department of Child Psychiatry evaluated through a questionnaire to be applied to their families.
  Interventions: Other: Not Applicable (observation)
- Healthy children: The orofacial trauma history, dietary habits and lifestyle changes of healthy children aged 3-14 years applying to Istanbul University Faculty of Dentistry Department of Pediatric Dentistry will be evaluated through a questionnaire to be applied to their families.
  Interventions: Other: Not Applicable (observation)

INTERVENTIONS:
Other: Not Applicable (observation) — Questionnaire

SUMMARY:
The Covid-19 outbreak has caused families and individuals to change their life routines and eating habits, and has affected their psychology, especially for children with autism, due to the change in their routines. These psychological changes may trigger the self-harming behavior that is very common in children with autism.

Dental trauma, a common problem in children and adolescents, can also be seen in individuals who need special care such as autism.

The aim of this study is to evaluate the susceptibility of children with autism to orofacial trauma during the pandemic period and compare them with the pre-pandemic period and the healthy group, as well as to question the lifestyle, nutritional habits, mood changes and oral health behaviors that may be related to the risk of trauma.

DETAILED DESCRIPTION:
The study is being carried out in Istanbul University Department of Pediatric Dentistry, period between September 2021 - March 2022 following the ethics committee approval 2021/49. Patient parents are informed about the study following the initial dental examination of the patient and the written informed consents are obtained from parents of all participants included in the study.

The orofacial trauma history, dietary habits and lifestyle changes of children aged 3-14 years diagnosed with autism in Istanbul University Department of Child Psychiatry and healthy children applying to Istanbul University Faculty of Dentistry Department of Pediatric Dentistry will be evaluated through a questionnaire to be applied to their families.

Questionnaire;

* 13 questions to question the sociodemographic profile,
* 10 questions to question the child's systemic disease history, oral hygiene habits and oral health status,
* 12 questions to question eating habits,
* 6 questions to question the child's lifestyle and psychological changes due to the Covid-19 pandemic,
* 20 questions to question the trauma story,
* In order to measure the DMFT/dmft status, 1 index will be filled and applied. Intraoral examinations of the children with autism who accepted to participate in the study, who came to the Istanbul University Child Psychiatry Department for examination, will also be examined, if there is any sign or history of trauma, it will be recorded and the possible causes of the trauma, its type, time, place and accompanying clinical findings will be evaluated and risk factors that may cause trauma (overjet/overbite) will be recorded.
* While evaluating dental traumas, hard tissue and periodontal tissue injuries will be recorded separately.
* Since X-rays cannot be taken from these patients, traumas related to the root in hard tissue injuries will not be evaluated.
* The amount of overjet and overbite; will be examined using an intraoral mirror and a periodontal probe. The amount of overjet will be recorded by measuring the distance of the upper incisors to the lower incisors when the jaws are in normal closing. When measuring the amount of overbite, the amount of covering the cutting edges of the lower incisors by the cutting edges of the upper incisors will be determined when the jaws are in normal closing.
* In addition, the patients with autism who came to the Department of Child Psychiatry of Istanbul University for examination and who accepted to participate in the study, will be measured with the help of the DMFT/dmft index, whether they have a history of trauma or not, while performing intraoral examinations.

A control group will be formed from healthy children who applied to the Pediatric Dentistry Department of Istanbul University without autism, taking into account the gender and age distribution of children with autism. Then, the groups will be compared within themselves and with each other, taking into account the pandemic period and before.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Children between the ages of 3-14 who have been diagnosed with autism
* Healthy children aged 3-14 years
* Presence of parents who can adequately answer the questionnaire questions

Exclusion Criteria:

* Not willing to participate in the study
* Patients with an unclear diagnosis of autism
* Those younger than 3 years old and over 14 years old
* In case of not being able to answer the questionnaire questions from the parents or remembering the trauma history

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 200 patients per month in the 3-14 age group who are being followed up with a diagnosis of autism from the Department of Child Psychiatry of Istanbul University, and 165 children will be selected by simple random sampling method from among the patients who applied to the clinic during the study period. On the other hand, healthy controls who applied to Istanbul University Faculty of Dentistry, Department of Pedodontics between September 6, 2021 and March 31, 2022 and met the inclusion criteria will be included in the order of application to the outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of the COVID-19 pandemic | 1 year
  The orofacial trauma history, dietary habits and lifestyle changes of children aged 3-14 years diagnosed with autism in Istanbul University Department of Child Psychiatry and healthy children applying to Istanbul University Faculty of Dentistry Department of Pediatric Dentistry will be evaluated through a questionnaire to be applied to their families.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Pinar Erdem, Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No